CLINICAL TRIAL: NCT05778656
Title: Cardiovascular Risk Prevention With a Mediterranean Dietary Pattern Reduced in Saturated Fat (CADIMED): Randomized Controlled Dietary Intervention Study With Metabolomic and Gut Microbiome Analyses
Brief Title: Cardiovascular Risk Prevention With a Mediterranean Dietary Pattern Reduced in Saturated Fat
Acronym: CADIMED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Granada (Other)
Collaborators: University of Oxford (Other); University of Copenhagen (Other); Norwegian Veterinary Institute (Unknown); Harvard University (Other); University Hospital Virgen de las Nieves (Other)
Responsible Party: Principal Investigator, Carmen Piernas Sanchez, Senior researcher, Universidad de Granada
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CADIMED2022
Record Dates: First submitted 2023-02-06; First posted 2023-03-21 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: LDL Cholesterol
Keywords: cardiovascular disease; Mediterranean diet; saturated fat; LDL cholesterol; red meat; fatty acids
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Fatty Acids

STUDY DESIGN:
Intervention Model Description: The CADIMED study is a randomized, controlled nutritional intervention study (two-arm parallel group design with a 1:1 ratio)
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: A computer-generated randomization with a stratified block design will be used, with sex, age, obesity, and fiber intake as stratification variables using randomly permuted blocks of size 2 and 4. The computer program (RedCap) will reveal the group allocation to the researcher, with no option to visualize the groups that will be assigned to future patients.
  It will not be possible to blind patients to the intervention group due to the nature of the intervention. However, the effectiveness measure comparing trial arms (primary outcomes) are objectively measured outcomes (blood lipids and metabolites) and not subject to interpretation by researchers, limiting the effect that researcher knowledge of the intervention group could have on outcomes. Where possible, the study team taking all the outcome measurements will remain blind to group allocation throughout the trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mediterranean diet without red and/or processed meat (Experimental): They will receive motivation and behavioral support through a study specific website which will be accessed after randomization. The research team will give participants further information on the use of this website. One of the features of the website will allow participants to collect and self-monitor their dietary intakes using 24h dietary recalls. Participants will be instructed to fill in as many recalls as possible throughout the study, with a minimum of 2 recalls at baseline and 2 recalls at follow up. Other features of the website include specific indications to eliminate red and processed meat in the context of a healthy Mediterranean dietary pattern, considering the key elements proposed in the dietary guidelines to improve cardiovascular health. The website will also provide them general information about the Mediterranean diet, as well as recipes, tips, and alternatives to replace meat when cooking at home or eating out. The rest of the clinical care will be as usual.
  Interventions: Behavioral: Cardiovascular Risk Prevention with a Mediterranean Dietary Pattern Reduced in Saturated Fat
- General advice based on the Mediterranean diet (No Intervention): The control group will be guided to use the same website although they will only have access to a restricted version of it, with the dietary recall feature plus general information about the Mediterranean diet. They will not receive specific recommendations to reduce red and processed meat or any other support or advice. Participants will be instructed to fill in as many 24h dietary recalls as possible throughout the study, with a minimum of 2 recalls at baseline and 2 recalls at follow up. The rest of the clinical care will be as usual.

INTERVENTIONS:
Behavioral: Cardiovascular Risk Prevention with a Mediterranean Dietary Pattern Reduced in Saturated Fat — Eight-week behavioral intervention consisting of a Mediterranean dietary pattern with elimination of red and processed meat
  Other Names: CADIMED
  Arms: Mediterranean diet without red and/or processed meat

SUMMARY:
The Cardiovascular Risk Prevention With a Mediterranean Dietary Pattern Reduced in Saturated Fat (CADIMED) study is a randomized, controlled intervention trial aiming to develop a dietary intervention that promotes saturated fat (SFA) reduction through eliminating red and processed meat consumption and to evaluate its impact on lipid and cardiovascular disease (CVD) risk biomarkers.

The main research question is:

* Does lowering SFA intake from specific foods (e.g., red and processed meat) modify cardiovascular risk factors in a Mediterranean dietary pattern context?

The aim is to compare, in a sample of 156 adult subjects (>18 years) with dyslipidemia, the effect of an intervention that promotes the elimination of red and processed meat intake vs. the control group that will follow the usual health advice for CVD prevention. Changes in CVD risk biomarkers, blood metabolomics and the microbiome will be investigated after 8 weeks of intervention.

DETAILED DESCRIPTION:
1. BACKGROUND

   Globally, cardiovascular diseases (CVD) are the leading cause of mortality. The World Health Organization estimates that, in 2019, 32% of deaths worldwide were due to CVD, mainly acute myocardial infarction. The most important cardiovascular risk factors are modifiable and are associated with poor diet, lack of physical activity, tobacco and alcohol consumption. Among them, it has been shown that an adequate diet is essential for the prevention of CVD given its effects on blood pressure, lipids, obesity, inflammation and endothelial function Amongst all dietary risk factors, saturated fatty acids (SFA) are of great interest because of their effects on low-density lipoprotein cholesterol (LDL-C) and total cholesterol, which are associated with increased cardiovascular risk due to endothelial dysfunction and atherosclerosis. Because of this, different organizations and institutions, such as the American Heart Association and the European Society of Cardiology, advise that SFA should represent less than 10% of total energy intake, preferably between 5% and 6% to prevent CVD. A Cochrane meta-analysis of clinical trials has shown that reducing SFA consumption decreases LDL-C significantly and up to 17% of cardiovascular events.

   Current clinical practice guidelines on the prevention and treatment of CVD generally recommend a low-SFA healthy diet but do not offer detailed or specific advice for effective interventions. This is important as different food sources of SFA may have different health risks. Foods contain complex mixtures of SFA, and evidence suggests that some fatty acids, such as lauric, myristic, and palmitic acid, may pose different risks. In particular, red meat contains a high proportion of palmitic acid [long-chain SFA (16:0)] and, although the current evidence is inconsistent and mainly based on observational studies, an increased risk of CVD has been associated with a higher intake of red and processed meat compared to plant protein sources, probably mediated by changes in lipid profile, inflammation or insulin resistance. However, other SFA-rich foods, such as milk and cheese, contain high proportions of shorter-chain fatty acids [lauric (12:0) and myristic (14:0)] and have not shown an association with CVD. It has been suggested that dairy products have other elements, such as calcium, which may counteract the unfavorable physiological effects of SFA.

   The principal investigator of this project has recently conducted an intervention study to reduce dietary SFA in a population at cardiovascular risk, which found a non-significant decrease in SFA intake. However, beneficial changes in blood lipid profile were observed among those participants who reduced their consumption of red and processed meats the most, compared to those who reduced other sources of SFA as dairy. In general, the current evidence is limited but suggests that different sources of SFA and individual proportions of SFA in red and processed meat may influence the cardiovascular profile differently; therefore robust intervention studies are required to confirm this. Also, changes in the fatty acid and blood lipid profile resulting from a dietary approach based on a Mediterranean dietary pattern without red and processed meat are widely unknown. It is relevant to investigate how these dietary modifications affect cardiovascular risk factors in the context of a Mediterranean diet in which consumption of unsaturated fats from olive oil or nuts confers benefits for CVD prevention.

   On the other hand, despite recent public health efforts, the reduction of SFA consumption through education or information programs in the population has not been sufficient. Previous research has established that it is possible to reduce the intake of SFA-rich foods by providing foods that replace them, and/or through intensive and adapted eating advice, requiring specialized staff and behavioral support. However, there is limited evidence on the effectiveness of less intensive and lower-cost interventions that can reach a greater number of people and have a significant effect on the population. Simple dietary guidelines that target specific foods (e.g., red meat) that are related to cardiovascular risk may have a greater potential to be adopted by an increasing number of people who need help to improve their diet quality and thus decrease their cardiovascular risk.

   The Cardiovascular Risk Prevention With a Mediterranean Dietary Pattern Reduced in Saturated Fat (CADIMED) study is a randomized, controlled intervention trial aiming to develop a dietary intervention that promotes saturated fat (SFA) reduction through eliminating red and processed meat consumption and to evaluate its impact on lipid and cardiometabolic biomarkers. The determination of lipid profiles, metabolomics, and gut microbiome will allow a better understanding of the questions raised and will help to establish simple dietary guidelines based on an effective approach for the treatment of dyslipidemia and prevention of CVD. All of this will be relevant to the third Sustainable Development Goal (SDG) of the United Nations Development Programme. The low cost and scalability of the intervention can help the Spanish healthcare system, particularly primary care, by helping to manage patients at risk of CVD and reduce healthcare costs. In addition, decreasing the consumption of red and processed meat also implies effects on global warming and environmental sustainability, contributing to achieving the 12th SDG.
2. OBJECTIVES

   Main objective:

   To develop a dietary intervention that promotes SFA reduction through eliminating red and processed meat consumption and to evaluate its impact on lipid and cardiovascular risk markers in adult patients with dyslipidemia.

   Specific objectives:
   1. To develop the necessary elements for the implementation of a dietary intervention that promotes the elimination of red and processed meats in adult patients with dyslipidemia.
   2. To test the effectiveness of a dietary approach that eliminates red and processed meat, in the context of a Mediterranean dietary pattern, on LDL-C and palmitic acid (main outcomes) after eight weeks of intervention, compared to the usual approach consisting of recommendations for a healthier lifestyle.
   3. To determine the metabolic alterations that occur in parallel with changes in SFA intake from red and processed meat, through a complete lipid and metabolomic profile, as well as the determination of other intermediate biomarkers of CVD.
   4. To evaluate the effect of the intervention on dietary intake and other lifestyle factors.
   5. To assess the effect of the intervention on the composition of the gut microbiota and its derived plasma metabolites.
   6. To establish a working panel of patients and members of the public (PPI) as well as health care professionals to improve the conduct, planing and management of the research as well as the dissemination of project results.
3. PROCEDURES AND DATA COLLECTION

The CADIMED study is a randomized, controlled nutritional intervention study (two-arm parallel group design), which will evaluate the effect of an eight-week behavioral intervention consisting of a Mediterranean eating pattern with elimination of red and processed meat, compared to the general advice for decreasing SFA intake in patients with high LDL-C. For this purpose, 156 patients, aged ≥ 18 years, with dyslipidemia and expressed desire to improve their diet and reduce CVD risk will be recruited.

3.1. Recruitment and pre-selection of patients

Recruitment for the CADIMED study will be conducted through healthcare professionals in primary or secondary care centers in Granada (Spain), who will help distribute information for participating in the study. Additionally, participants will be recruited from the community through posters and brochures displayed in doctors' offices and public spaces near healthcare facilities as well as adverts in social media and news outlets. Interested participants will be offered further information through the CADIMED website (www.cadimed.es) as well as details to contact the research team by phone, email or online questionnaire to confirm that they meet the essential inclusion criteria. An initial pre-screening questionnaire will be administered by phone and volunteers who meet the inclusion criteria will be scheduled for an initial visit with the research and clinical teams at Hospital Doctor Olóriz, Granada.

3.2. Informed consent

During the initial visit with the research team, study information will be given to patients (Patient Information Sheet and Informed Consent Form), and the informed consent form will be read and signed. Patients will have the chance to ask questions regarding the study and participation, and those who complete the informed consent form will be enrolled.

3.3. Questionnaires and measurements

The research team will administer a questionnaire to collect the patient's demographic characteristics, including age, sex, education, socioeconomic class, alcohol intake, physical activity, diet, and smoking, using an electronic data capture database (RedCap). The clinical team from Virgen de las Nieves Hospital will be responsible for registering the clinical data related to the medical history and/or use of drugs. Height, weight, and blood pressure will be measured following a standardized protocol, at baseline and follow up. A study website (designed especially to deliver the intervention) will be also used to collect dietary data through 24h recalls. This website will include each patient's unique code and an embedded diet questionnaire that should be completed at least twice a week during the first and last week of the intervention to obtain valid measures of usual intake. In addition, a food frequency questionnaire covering the previous 4 weeks will be also completed at baseline and follow up to assess the eating pattern.

3.4. Blood samples

Blood samples will be taken by the clinical team during the initial visit and at the end of the follow-up, after 8h of overnight fasting. These samples will be processed in the laboratory of Virgen de las Nieves Hospital for subsequent analysis in the hospital. Part of the samples will be transferred and analysed at the Institute of Nutrition and Food Technology (INYTA) laboratory.

3.5. Stool samples

Stool samples will be taken at the beginning and at the end of the follow-up. Patients will be provided with the necessary material and instructions for collection and storage of the samples. The samples will be processed for analysis at the INYTA laboratory.

3.6. Randomization and blinding

Once it is confirmed that the participant meets all the inclusion criteria, the intervention group will be randomly assigned and participants will receive the corresponding explanation regarding the intervention they get allocated to.

A computer-generated randomization with stratified block design will be used, with sex, age, obesity, and fiber intake as stratification variables using randomly permuted block sizes of 2 and 4. The computer program will reveal the allocation group to the researcher, with no option to visualize the groups that will be assigned to future patients.

It will not be possible to blind patients to the intervention group due to the nature of the intervention. However, the effectiveness measures (primary outcomes) are objectively measured outcomes (blood lipids and metabolites) which means they are not subject to interpretation by researchers, limiting the effect that researcher knowledge of the intervention group could have on outcomes. Where possible, the study team taking all the outcome measurements will remain blind to group allocation throughout the trial. Participants will only be aware of the trial arm that they are exposed to and will be unaware of the other trial arm.

3.7. Discontinuation/Withdrawal and End of Study

Participants will be informed that they have the right to withdraw from the study at any time. Participants that are withdrawn or discontinued/lost to follow up will not be replaced as a sufficient sample size will be recruited to allow for non-completion rate. Participants will be asked to consent for the use of their data up to the point of discontinuation/lost to follow up.

The end of study will be completed after all the follow up questionnaires and measurements are taken.

3.8. Statistical analysis

1. Sample size: a recent randomized controlled trial in a UK adult population with dyslipidemia, in which similar dietary approaches for reducing SFA intake were tested, showed a change in LDL-C of approximately 15 mg/dl (SD26) in the intervention group that achieved a greater reduction in meat intake (14). If 78 participants are recruited in each group (n = 156), it will be possible to detect a minimum difference of 15 mg/dl between the intervention and control group, with 90% power, two-sided α = 0.05 and accounting for 20% attrition rate using intention-to-treat analysis.
2. Statistical analysis of primary and secondary outcomes: baseline characteristics will be summarized using descriptive statistics by trial arm. Statistical analysis will be performed with STATA IC 16.0 software (College Station, TX: StataCorp LLC 2019). Descriptive statistics will be reported with standard deviation (SD) and 95% confidence intervals. Continuous variables will be presented as mean and SD unless the use of the median and interquartile range is needed. Categorical variables will be expressed as frequencies and percentages. The effectiveness outcomes will be analyzed on an intention-to-treat basis, that is, all participants will be analyzed according to the group to which they were randomly allocated, regardless of their compliance. Analysis of effectiveness measures will use data from all participants for whom a baseline and follow-up measure exist. A linear regression model will be used to calculate the difference of means with 95% confidence intervals, with adjustment for baseline levels of the dependent variable and recruitment site. Before the analysis, the assumptions of linear regression, specifically homoscedasticity, and the normality of the distribution of residuals will be explored. Where these assumptions are not met, suitable non-parametric analyses will be employed. The sensitivity of the results to confounding due to differences in baseline characteristics will be also examined; as well as the sensitivity of imputing missing outcome data using baseline-observation carried forwards (using the baseline value) and multiple imputation (using group allocation and patient's characteristics to impute the missing data). An exploratory subgroups analysis of outcomes by sociodemographic characteristics will be performed.

3.9. Assessment of metabolomic profiles and gut microbiota

This project will employ a metabolomic and metagenomic profiling approach (gut microbiota) using state-of-the-art analytical technologies to provide deeper understanding of the metabolic responses to the proposed dietary intervention (elimination of red/processed meat intake) in the context of a Mediterranean dietary pattern. Lipid profiling and a complete metabolomic and metagenomic analysis will be performed to investigate specific changes observed in intervention group compared to control. These assessments will be performed at the at the Institute of Nutrition and Food Technology (INYTA) or third-party laboratories where needed. Once the main assessments have been carried out and with prior consent, the surplus of these samples with their corresponding code will be stored at -80ºC in the Public Health System of Andalusian Biobank (PHSABB), for further analysis related to the project, including aliquots with leukocytes for DNA extraction and erythrocytes for studies of antioxidant defense enzymes.

3.10. Ethical and legal considerations

The study team will ensure that this study is conducted in accordance with the principles of the Declaration of Helsinki.

The protocol, informed consent form and participant information sheet was approved by the ethical committee: "Comité de Ética de Investigación Biomédica de la Provincia de Granada" (CEI/CEIM Granada). Date of approval 30/11/2022; Study code 1831-N-22

Funding for this study is provided by:

* Ministry of Science and Innovation, Knowledge Generation Projects 2021, PID2021-127312OA-I00
* Ministry of Science and Innovation, Ramon y Cajal 2020 call, RYC2020-028818-I,

All data collected from patients will be stored in a password-protected database and encoded/anonymised with a unique code for each patient (RedCap). Only the research team and the health authorities, who have the duty to keep confidentiality, will have access to all the data collected for the study. Only information that cannot be identified may be transmitted to third parties.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form.
* Age ≥18 years to ≤75 years.
* With indication to start lifestyle intervention based on recent values (e.g., last 3-6 months) of LDL-C ≥ 116 mg/dl and < 190 mg/dl; or as long as pharmacological treatment has not been advised and started (ESC/EAS Guide, Rev Esp Cardiol. 2020).
* Access to a device (e.g., smartphone, tablet, computer) with internet and digital skills to use the website.
* Motivation and willingness to be assigned to any group to improve their diet and commitment to perform the designated protocol.

Exclusion Criteria:

* Patients with familial hypercholesterolemia and/or on treatment with lipid-lowering drugs (including statins, ezetimibe, PCSK9 inhibitors, fibrates, bile acid sequestrants, omega-3 fatty acids, nicotinic acid/Vit B3), dietary supplements or functional foods for the treatment of dyslipidemia (plant sterols, monacolin, red yeast rice, fiber supplements 3-10 g (Plantago), policosanol, berberine, and soy protein/lecithin) in the last 3 months.
* High cardiovascular risk that requires pharmacological treatment, for example, patients with recent and/or established CVD, type 1 and 2 diabetes.
* Uncompensated thyroid function disorders; relevant comorbidities (including liver failure and cholestasis, chronic kidney disease, Cushing's syndrome, nephrotic syndrome, class III obesity - BMI ≥ 40 kg/m²); cancer; psychiatric disorders and/or that in the opinion of the investigator hinder the fulfillment or follow-up of the study.
* Excessive alcohol consumption: > 40 g/d (4 UBEs/day) in men and > 20-25 g/d (2-2.5 UBEs/day) in women (Ministry of Health, July 2020).
* Pregnancy, lactation, perimenopause (amenorrhea < 1 year) and women who change, start, or finish their treatment with hormonal contraceptives during the study.
* Enrollment in other research studies or following restricted eating patterns (e.g., vegetarians and vegans) that could interfere with study requirements.
* Failure to grant informed consent or not complete the initial assessment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 157 (Actual)
Dates: Start 2023-03-19 (Actual); Primary Completion 2025-08-06 (Actual); Study Completion 2025-08-06 (Actual)

PRIMARY OUTCOMES:
LDL-Cholesterol (mg/dL) | 8 weeks
  To investigate changes in LDL-C after 8 weeks in the intervention group compared to control
Fatty acid profile (%) | 8 weeks
  The initial plan was to investigate changes in palmitic acid after 8 weeks in the intervention group compared to control. However, after careful consideration with experts in Biochemistry, it is proposed to measure the overall fatty acid profile in erytrocyte membranes (instead of measuring palmitic acid individually for the primary outcome and the rest of individual fatty acids for the secondary outcome measures). Given the nature of this dietary intervention and the homeostatic metabolic processes that regulate individual fatty acids, it is advised to look at changes in the overall fatty acid profile (ie. their relative proportion within the overall profile) in response to the intervention. This change does not affect any methodological aspect of the trial because the sample size was calculated based on the primary outcome LDL-cholesterol change (see Statistical Analysis in Study Description)

SECONDARY OUTCOMES:
Metabolites derived from lipid and metabolomic profile analysis (mg/dL) | 8 weeks
  To investigate changes in other circulating biomarkers such as HDL-C, total cholesterol, triglycerides, and endogenous and exogenous metabolites related to CVD risk and meat consumption (all expressed as mg/dL) after 8 weeks in the intervention group compared to control.
Metabolites derived from lipid and metabolomic profile analysis (percentage) | 8 weeks
  To investigate changes in other circulating biomarkers such as HDL-C, non-HDL-C, total cholesterol, triglycerides, and endogenous and exogenous metabolites related to CVD risk and meat consumption (all expressed as percentages) after 8 weeks in the intervention group compared to control.
CVD risk related markers: C-reactive protein, IL-6, IL8/CXCL8, IL10, IL23, TNF-alpha, IFNgamma, ICAM1, VCAM1, ELAM1, MPO, endotelin I, angiotensin II (ng/mL) | 8 weeks
  To investigate changes in other biomarkers of inflammation and endothelial damage ( C-reactive protein, IL-6, IL8/CXCL8, IL10, IL23, TNF-alpha, IFNgamma, ICAM1, VCAM1, ELAM1, MPO, endotelin I, angiotensin II, all expressed as ng/mL) after 8 weeks in the intervention group compared to control.
CVD risk related markers: Glucose (mg/dL) | 8 weeks
  To investigate changes in other biomarkers of insulin resistance and diabetes: glucose (mg/dL) after 8 weeks in the intervention group compared to control.
CVD risk related markers: Insulin (mU/ml) | 8 weeks
  To investigate changes in other biomarkers of insulin resistance and diabetes: insulin (mU/ml) after 8 weeks in the intervention group compared to control.
CVD risk related markers: HbA1c (percentage) | 8 weeks
  To investigate changes in other biomarkers of insulin resistance and diabetes: HbA1c (percentage) after 8 weeks in the intervention group compared to control.
CVD risk related markers: systolic and diastolic blood pressure (mmHg) | 8 weeks
  To investigate changes in sistolic and diastolic blood pressure (mmHg) after 8 weeks in the intervention group compared to control.
CVD risk related markers: weight (kg) | 8 weeks
  To investigate changes in weight (kg) and body mass index (calculated as the weight in kg divided by the squared height in m) after 8 weeks in the intervention group compared to control.
CVD risk related markers: waist circumference (cm) | 8 weeks
  To investigate changes in waist circumference (cm) after 8 weeks in the intervention group compared to control.
Gut microbiome composition | 8 weeks
  To investigate changes in the gut microbiome composition (percentage of each species) after 8 weeks in the intervention group compared to control.
Gut microbiome derived metabolites | 8 weeks
  To investigate changes in the gut microbiome derived metabolites: Lipopolysaccharides (LPS), Lipoprotein binding LPS and other relevant microbiome metabolites (all measured in microgram/mL) after 8 weeks in the intervention group compared to control.
Dietary intake: total daily energy intake (kcal) | 8 weeks
  To investigate changes in total daily energy intake (kcal) after 8 weeks in the intervention group compared to control.
Dietary intake: meat consumption (gr) | 8 weeks
  To investigate changes in red and processed meat consumption per day (gr) after 8 weeks in the intervention group compared to control.
Dietary intake: meat consumption (kcal) | 8 weeks
  To investigate changes in red and processed meat consumption per day (kcal) after 8 weeks in the intervention group compared to control.
Dietary intake: meat consumption (percentage of energy intake) | 8 weeks
  To investigate changes in red and processed meat consumption per day (percentage of energy intake) after 8 weeks in the intervention group compared to control.
Dietary intake: relevant macro and micronutrients (gr) | 8 weeks
  To investigate changes in total daily intake of macro- and micronutrients: saturated fatty acids, total fat, total sugars, total carbohydrates, total protein, fiber, salt (all expressed in gr) after 8 weeks in the intervention group compared to control.
Dietary intake: relevant macro and micronutrients (kcal) | 8 weeks
  To investigate changes in total daily intake of macro- and micronutrients: saturated fatty acids, total fat, total sugars, total carbohydrates, total protein, fiber, salt (all expressed in kcal) after 8 weeks in the intervention group compared to control.
Dietary intake: relevant macro and micronutrients (percentage of energy) | 8 weeks
  To investigate changes in total daily intake of macro- and micronutrients: saturated fatty acids, total fat, total sugars, total carbohydrates, total protein, fiber, salt (all expressed in percentage of energy intake) after 8 weeks in the intervention group compared to control.
Dietary intake: dietary patterns (z score) | 8 weeks
  To investigate changes in general dietary patterns (combinations of individual food group intakes, expressed as a z score which negative values indicate low adherence and positive values indicate high adherence) after 8 weeks in the intervention group compared to control.
Other lifestyle factors: physical activity (minutes) | 8 weeks
  To investigate changes in physical activity (minutes of moderate or vigorous PA per day) after 8 weeks in the intervention group compared to control.
Other lifestyle factors: smoking (cigerettes/day) | 8 weeks
  To investigate changes in smoking (cigarettes per day) after 8 weeks in the intervention group compared to control.
Other lifestyle factors: alcohol intake (units/day) | 8 weeks
  To investigate changes in alcohol intake (units/day) after 8 weeks in the intervention group compared to control.

OTHER OUTCOMES:
Process Evaluation Outcomes: feasibility outcomes | 8 weeks
  Process evaluation analysis of quantitative and qualitative measures to understand why and how the the intervention was effective. The following feasibility outcomes will be explored: the rate of volunteer recruitment (%), eligible (%) and the rate of patients completing the study (%)
Process Evaluation Outcomes: acceptance and use of the intervention | 8 weeks
  Process evaluation analysis of quantitative and qualitative measures to understand why and how the the intervention was effective. Measures of acceptance of the intervention, app use, knowledge about diet and cardiovascular disease and evidence of contamination of the control group will be collected through questionnaires at the end of follow-up. Descriptive analyses will be performed using the answers to these questions (scales 1-5, 1 indicating low acceptance and 5 indicating high acceptance).
Exploratory subgroup analyses by SES | 8 weeks
  An exploratory subgroups analysis of outcomes by sociodemographic characteristics (age group, sex, education/income group) will be performed

CONTACTS AND LOCATIONS:
Overall Officials: Carmen Piernas, PhD, Principal Investigator — Universidad de Granada
Locations (1):
- University of Granada, Granada, Granada, Spain

IPD SHARING:
Plan to Share IPD: Undecided
A data sharing plan will be drafted after study closure and before data analysis

REFERENCES:
- [Background] World Health Organization. Cardiovascular diseases (CVDs). WHO: Copenhagen; 2021. Available in: https://www.who.int/news-room/fact-sheets/detail/cardiovascular-diseases-(cvds)
- [Background] Verschuren WMM, Boer JMA, Temme EHM. Optimal diet for cardiovascular and planetary health. Heart. 2022 Jul 13;108(15):1234-1239. doi: 10.1136/heartjnl-2019-316373. No abstract available. PMID 34635484
- [Background] Davignon J, Ganz P. Role of endothelial dysfunction in atherosclerosis. Circulation. 2004 Jun 15;109(23 Suppl 1):III27-32. doi: 10.1161/01.CIR.0000131515.03336.f8. PMID 15198963
- [Background] SEC Working Group for the 2021 ESC guidelines on cardiovascular disease prevention in clinical practice and SEC Guidelines Committee. Comments on the 2021 ESC guidelines on cardiovascular disease prevention in clinical practice. Rev Esp Cardiol (Engl Ed). 2022 May;75(5):364-369. doi: 10.1016/j.rec.2021.10.023. Epub 2022 Feb 11. No abstract available. English, Spanish. PMID 35165071
- [Background] American Heart Association. Saturated Fat. AHA: Texas: 2021. Available in: https://www.heart.org/en/healthy-living/healthy-eating/eat-smart/fats/saturated-fats
- [Background] Hooper L, Martin N, Jimoh OF, Kirk C, Foster E, Abdelhamid AS. Reduction in saturated fat intake for cardiovascular disease. Cochrane Database Syst Rev. 2020 Aug 21;8(8):CD011737. doi: 10.1002/14651858.CD011737.pub3. PMID 32827219
- [Background] Astrup A, Magkos F, Bier DM, Brenna JT, de Oliveira Otto MC, Hill JO, King JC, Mente A, Ordovas JM, Volek JS, Yusuf S, Krauss RM. Saturated Fats and Health: A Reassessment and Proposal for Food-Based Recommendations: JACC State-of-the-Art Review. J Am Coll Cardiol. 2020 Aug 18;76(7):844-857. doi: 10.1016/j.jacc.2020.05.077. Epub 2020 Jun 17. PMID 32562735
- [Background] Chowdhury R, Warnakula S, Kunutsor S, Crowe F, Ward HA, Johnson L, Franco OH, Butterworth AS, Forouhi NG, Thompson SG, Khaw KT, Mozaffarian D, Danesh J, Di Angelantonio E. Association of dietary, circulating, and supplement fatty acids with coronary risk: a systematic review and meta-analysis. Ann Intern Med. 2014 Mar 18;160(6):398-406. doi: 10.7326/M13-1788. PMID 24723079
- [Background] Zong G, Li Y, Wanders AJ, Alssema M, Zock PL, Willett WC, Hu FB, Sun Q. Intake of individual saturated fatty acids and risk of coronary heart disease in US men and women: two prospective longitudinal cohort studies. BMJ. 2016 Nov 23;355:i5796. doi: 10.1136/bmj.i5796. PMID 27881409
- [Background] Guasch-Ferre M, Satija A, Blondin SA, Janiszewski M, Emlen E, O'Connor LE, Campbell WW, Hu FB, Willett WC, Stampfer MJ. Meta-Analysis of Randomized Controlled Trials of Red Meat Consumption in Comparison With Various Comparison Diets on Cardiovascular Risk Factors. Circulation. 2019 Apr 9;139(15):1828-1845. doi: 10.1161/CIRCULATIONAHA.118.035225. PMID 30958719
- [Background] Key TJ, Appleby PN, Bradbury KE, Sweeting M, Wood A, Johansson I, Kuhn T, Steur M, Weiderpass E, Wennberg M, Lund Wurtz AM, Agudo A, Andersson J, Arriola L, Boeing H, Boer JMA, Bonnet F, Boutron-Ruault MC, Cross AJ, Ericson U, Fagherazzi G, Ferrari P, Gunter M, Huerta JM, Katzke V, Khaw KT, Krogh V, La Vecchia C, Matullo G, Moreno-Iribas C, Naska A, Nilsson LM, Olsen A, Overvad K, Palli D, Panico S, Molina-Portillo E, Quiros JR, Skeie G, Sluijs I, Sonestedt E, Stepien M, Tjonneland A, Trichopoulou A, Tumino R, Tzoulaki I, van der Schouw YT, Verschuren WMM, di Angelantonio E, Langenberg C, Forouhi N, Wareham N, Butterworth A, Riboli E, Danesh J. Consumption of Meat, Fish, Dairy Products, and Eggs and Risk of Ischemic Heart Disease. Circulation. 2019 Jun 18;139(25):2835-2845. doi: 10.1161/CIRCULATIONAHA.118.038813. Epub 2019 Apr 22. PMID 31006335
- [Background] Visioli F, Poli A. Fatty Acids and Cardiovascular Risk. Evidence, Lack of Evidence, and Diligence. Nutrients. 2020 Dec 9;12(12):3782. doi: 10.3390/nu12123782. PMID 33317164
- [Background] de Oliveira Otto MC, Mozaffarian D, Kromhout D, Bertoni AG, Sibley CT, Jacobs DR Jr, Nettleton JA. Dietary intake of saturated fat by food source and incident cardiovascular disease: the Multi-Ethnic Study of Atherosclerosis. Am J Clin Nutr. 2012 Aug;96(2):397-404. doi: 10.3945/ajcn.112.037770. Epub 2012 Jul 3. PMID 22760560
- [Background] Piernas C, Aveyard P, Lee C, Tsiountsioura M, Noreik M, Astbury NM, Oke J, Madigan C, Jebb SA. Evaluation of an intervention to provide brief support and personalized feedback on food shopping to reduce saturated fat intake (PC-SHOP): A randomized controlled trial. PLoS Med. 2020 Nov 5;17(11):e1003385. doi: 10.1371/journal.pmed.1003385. eCollection 2020 Nov. PMID 33151934
- [Background] Estruch R, Ros E, Salas-Salvado J, Covas MI, Corella D, Aros F, Gomez-Gracia E, Ruiz-Gutierrez V, Fiol M, Lapetra J, Lamuela-Raventos RM, Serra-Majem L, Pinto X, Basora J, Munoz MA, Sorli JV, Martinez JA, Fito M, Gea A, Hernan MA, Martinez-Gonzalez MA; PREDIMED Study Investigators. Primary Prevention of Cardiovascular Disease with a Mediterranean Diet Supplemented with Extra-Virgin Olive Oil or Nuts. N Engl J Med. 2018 Jun 21;378(25):e34. doi: 10.1056/NEJMoa1800389. Epub 2018 Jun 13. PMID 29897866
- [Background] Reidlinger DP, Darzi J, Hall WL, Seed PT, Chowienczyk PJ, Sanders TA; Cardiovascular disease risk REduction Study (CRESSIDA) investigators. How effective are current dietary guidelines for cardiovascular disease prevention in healthy middle-aged and older men and women? A randomized controlled trial. Am J Clin Nutr. 2015 May;101(5):922-30. doi: 10.3945/ajcn.114.097352. Epub 2015 Mar 18. PMID 25787998
- [Background] Vafeiadou K, Weech M, Altowaijri H, Todd S, Yaqoob P, Jackson KG, Lovegrove JA. Replacement of saturated with unsaturated fats had no impact on vascular function but beneficial effects on lipid biomarkers, E-selectin, and blood pressure: results from the randomized, controlled Dietary Intervention and VAScular function (DIVAS) study. Am J Clin Nutr. 2015 Jul;102(1):40-8. doi: 10.3945/ajcn.114.097089. Epub 2015 May 27. PMID 26016869
- [Background] Lin JS, O'Connor E, Whitlock EP, Beil TL. Behavioral counseling to promote physical activity and a healthful diet to prevent cardiovascular disease in adults: a systematic review for the U.S. Preventive Services Task Force. Ann Intern Med. 2010 Dec 7;153(11):736-50. doi: 10.7326/0003-4819-153-11-201012070-00007. PMID 21135297
- [Derived] Chavez-Alfaro L, Tenorio Jimenez C, Silveira-Sanguino V, Noguera Gomez MJ, Fernandez-Moreno C, Rodriguez Cuesta AM, Lebron Arana AF, Segura Calvo O, Merino De Haro I, Aguilera CM, Gomez-Llorente C, Rangel-Huerta OD, Astbury N, Perez-Cornago A, Guasch-Ferre M, Piernas C. Intervention design and adherence to Mediterranean diet in the Cardiovascular Risk Prevention with a Mediterranean Dietary Pattern Reduced in Saturated Fat (CADIMED) randomized trial. Nutr Res. 2025 Apr;136:120-132. doi: 10.1016/j.nutres.2025.03.001. Epub 2025 Mar 10. PMID 40187224

DOCUMENTS (3):
  • Study Protocol and Informed Consent Form (2023-02-03): https://cdn.clinicaltrials.gov/large-docs/56/NCT05778656/Prot_ICF_001.pdf
  • Statistical Analysis Plan: SAP v2.0 (2025-12-18): https://cdn.clinicaltrials.gov/large-docs/56/NCT05778656/SAP_002.pdf
  • Statistical Analysis Plan: SAP v 1.0 (2025-07-16): https://cdn.clinicaltrials.gov/large-docs/56/NCT05778656/SAP_000.pdf